CLINICAL TRIAL: NCT05124704
Title: Propofol EC50 for Inducing Loss of Consciousness in Gastrectomy: Combined General and Epidural Anesthesia Versus General Anesthesia
Brief Title: Propofol EC50 for Inducing Loss of Consciousness in General Combined Epidural Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wang Jiangling (Other)
Responsible Party: Sponsor-Investigator, Wang Jiangling, Clinical Resident, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2021-214
Record Dates: First submitted 2021-10-11; First posted 2021-11-18 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer
Keywords: Propofol EC50; Epidural anesthesia; Gastric cancer; Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: 60 adult gastric cancer patients between 18-75 years, ASA physical state I and II, undergoing open gastrectomy, were enrolled in this study.
  Epidural puncture was performed in the left lateral position through the interspace between the eighth to ninth thoracic vertebra (T8-T9). Epidural catheter was inserted. In group TEA+GA, 5-8ml of 0.375% ropivacaine depend on the height and weight of the patient was administrated through the epidural catheter at least 20 min before induction, to obtain a bilateral segmentary sensory block to pinprick between T4 and T12 dermatomes. Continuous infusion of 4-6 ml 0.375% ropivacaine was applied using micro-infusion pump after induction. In group GA, same dose of normal saline was administered before induction and during surgery.
Who Masked: Participant, Investigator
Masking Description: Epidural puncture was performed by the fist anesthesiologist. First dosage and continuous infusion of ropivacaine was administered by the second anesthesiologist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined epidural with general anesthesia (Experimental): Patients in this group received 5-8ml of 0.375% ropivacaine depend on the height and weight of the patient was administrated through the epidural catheter at least 20 min before induction.Followed by a continuous infusion of 4-6 ml 0.375% ropivacaine was applied using micro-infusion pump after induction during surgery.
  Interventions: Drug: 5-8ml 0.375% ropivacaine
- General anesthesia (Sham Comparator): In this group, same dose of normal saline was administered before induction and during surgery.
  Interventions: Other: 5-8ml normal saline

INTERVENTIONS:
Drug: 5-8ml 0.375% ropivacaine — 5-8ml of 0.375% ropivacaine depend on the height and weight of the patient was administrated through the epidural catheter at least 20 min before induction in experimental group. Followed by a continuous infusion of 4-6 ml/h using micro-infusion pump after induction during surgery.
  Other Names: Experimental
  Arms: Combined epidural with general anesthesia
Other: 5-8ml normal saline — 5-8ml of normal saline depend on the height and weight of the patient was administrated through the epidural catheter at least 20 min before induction. Followed by a continuous infusion of 4-6 ml/h using micro-infusion pump after induction during surgery.
  Other Names: Sham control
  Arms: General anesthesia

SUMMARY:
The beneficial of perioperative usage of thoracic epidural anesthesia and analgesia in various thoracic and upper abdominal surgery are well studied. However, intraoperative data are lacking whether combined thoracic epidural and general anesthesia have effect on the median (50%) effective effect-concentration (EC50) of propofol for inducing loss of consciousness (LOC). We performed this study among patients undergoing open gastrectomy in gastric cancer patients.

Sixty patients undergoing open gastrectomy were randomly assigned to two groups with thoracic combined general anesthesia (TEA+GA) or general anesthesia (GA) alone. Target-controlled infusion (TCI) of propofol was used for anesthesia induction. The initial propofol concentration of target effect-site (Ceprop) was 3.5 ug/ml and was increased stepwise by 0.5ug/ml at each 4 min intervals by an un-down sequential method to reach LOC. The predicted Ceprop at the time of LOC, intravenous anesthetics, vasopressor requirement, emergency time from anesthesia and postoperative numeric rating scale (NRS) were recorded and analyzed between two groups.

DETAILED DESCRIPTION:
After received the approvement of ethics committee of the Cancer Hospital of the University of Chinese Academy of Sciences (approval number IRB- 2021-214). 60 adult gastric cancer patients between 18-75 yrs, ASA physical state I and II, undergoing open gastrectomy, were enrolled in this study. The exclusion criteria included: patients with contraindications to epidural puncture or catheter placement; chronic or acute (within 48 h) intake of psychotropic drugs, benzodiazepines, anticonvulsants, or opioids; alcoholism; hepatic, renal, neurological or other organ dysfunction; younger than 18 years or older than 75 years; with allergic to local anesthetic solutions or opioids; received neo-adjuvant chemotherapy; as well as patients who refuse to receive epidural puncture.

Patients were randomly assigned to either TEA+GA group of GA group. The requirement for the modified up-down method was used to confirm sample size (1).

Preoperative arrangements 3-lead electrocardiogram, pulse oximetry and continuously invasive artery blood pressure via left radial artery() were measured for basic monitoring. A central venous catheter was placed in the right internal jugular vein for fluid input and central venous pressure measurement and its position was confirmed by ultrasound. Bispectral Index (BIS) monitor (VT94306, Aspect VISTA, Covidien IIc, MA, USA) was measured for monitoring the depth of anesthetic.

Thoracic Epidural Anesthesia Epidural puncture was performed in the left lateral position through the interspace between the eighth to ninth thoracic vertebra (T8-T9). Epidural catheter was inserted by median approach using "loss-of-resistance"technique and was placed advanced 4 cm cephalad. A test dose of 3ml, 1%, lidocaine was injected through the catheter after the aspiration test for blood and cerebrospinal fluid shows negative results. Non sensory and motor anesthesia after 4 min of test dose injection indicate the absence of accidental subarachnoid placement of the catheter. In group TEA+GA, 5-8ml of 0.375% ropivacaine depend on the height and weight of the patient was administrated through the epidural catheter at least 20 min before induction, by the second anesthesiologist, to obtain a bilateral segmentary sensory block to pinprick between T4 and T12 dermatomes. Continuous infusion of 4-6 ml 0.375% ropivacaine was applied using micro-infusion pump after induction(2). In group GA, same dose of normal saline was administered before induction and during surgery.

General Anesthesia General anesthesia was induced by propofol plasma target-controlled infusion (TCI) (). To explore the EC50 of propofol for inducing LOC in two groups. We started induction using a series of predicted effect-site concentrations of propofol (Ceprop) with an equal step wise of 0.5 ug/ml, according to the up-down method of Dixon(1). The initial Ceprop for the first patient of each group was 3.5 ug/ml based on previous studies (3) . Positive response to propofol was defined as LOC happened within 4 min after start of TCI under initial concentration. Otherwise the response was taken as negative and propofol concentration was increased 0.5 ug/ml more each 4 min until patient reach LOC (LOC was defined as loss of response to verbal commands). The initial TCI Ceprop was increased by 0.5 ug/ml for the next patients if the previous patient shows negative in the same group. The initial TCI Ceprop was decreased by 0.5 ug/ml for the next patient if the previous patient shows positive in the same group. All the patients were increased by 0.5 ug/ml stepwise at 4 min intervals until they showed LOC. An interval of 4 min was based on the pharmacokinetic and pharmacodynamic (PK-PD) character of propofol in order to obtain the steady-state effect-site concentrations (4; 5). An intravenous of 0.25 mg/Kg oxycodone and 0.6 mg/Kg rocuronium were given after LOC to facilitate tracheal intubation.

Maintenance of anesthesia Anesthesia was maintained with propofol, remifentanil and rocuronium during surgery. Ceprop was adjusted in stepwise of 0.5 ug/ml to keep the BIS between 45 to 55 in two groups. The lowest Ceprop was 2.0 ug/ml to avoid intraoperative awareness. Concentration for remifentanil was between 0.05 ug/Kg/min and 0.25 ug/Kg/ min during surgery depend on the blood pressure. The maintenance doses of rocuronium was 0.15mg/Kg as required to maintain surgical paralysis (6). Patients with hypertension were treated with 10 mg urapidil or 5 mg diltiazem i.v and hypotension was treated initially by speeding Ringger's solution, infusion voluven, then decrease concentration of remifentanil by 0.05 ug/Kg/min until reach the lower limit of 0.05 ug/Kg/min and finally given 5mg ephedrine i.v. 80 ug phenylephrine or 1mg metaraminol were then given if hypotension was remaining.

Postoperative management Anesthetics were stopped when the final surgical suture was done and then 2-4mg/Kg of sugammadex was applied according to the train-of-four (TOF) ratio. The duration between the time of discontinuation of anesthetics and the time of spontaneous opening of eyes was defined as anesthesia emergency time. All patients received postoperative patient-controlled epidural analgesia (PCEA) 0f 0.175% ropivacaine with 0.7ug/ml sufentanil. The PCEA continuous infusion dose was 3-4 ml with patient-controlled bolus dose of 4-5ml depend on the height and weight of patient.

Patients were transferred to PACU after extubation and stay at least 60 min there. In PACU, pain intensity using numerical analogue score of 0-10, postoperative nausea, vomiting and times of hypotension were evaluated and recorded at 30min, 60min and the time leave PACU.

ELIGIBILITY:
Inclusion Criteria:

Gastric cancer patients age between 18-75 yrs;

ASA physical state I and II

Undergoing open gastrectomy

Exclusion Criteria:

With contraindications to epidural puncture or catheter placement

Chronic or acute (within 48 h) intake of psychotropic drugs, benzodiazepines, anticonvulsants, or opioids; alcoholism

Hepatic, renal, neurological or other organ dysfunctiony

Younger than 18 years or older than 75 years

Allergic to local anesthetic solutions or opioids

Received neo-adjuvant chemotherapy

Refuse to receive epidural puncture

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiangling Wang, M.D, Principal Investigator — Cancer Hospital of The University of Chinese Academy of Sciences
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Shen Y, Guo W, Zhang W, Cui X, Cai S, Chen X. Propofol EC50 for inducing loss of consciousness in patients under combined epidural-general anesthesia or general anesthesia alone: a randomized double-blind study. Front Med (Lausanne). 2023 Nov 6;10:1194077. doi: 10.3389/fmed.2023.1194077. eCollection 2023. PMID 38020175

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combined Epidural With General Anesthesia | General Anesthesia
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Epidural With General Anesthesia | General Anesthesia | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 21 | 39
  >=65 years | 12 | 9 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59.5 [52.75 to 69.25] | 62 [54 to 69] | 60.5 [53.5 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 16 | 21 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Propofol EC50 for Inducing Loss of Conciousness
Description: Recording propofol EC50 for inducing loss of conciousness between general with epidural anesthesia group and general group with propofol effect-site target-controlled infusion (TCI) system
Time Frame: From anesthesia induction to patient loss of consciousness, an average of 5 minutes.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Combined Epidural With General Anesthesia | General Anesthesia
Number analyzed (Participants) | 30 | 30
ug/ml | 2.97 (0.44) | 3.36 (0.22)

2. Primary Outcome: Predicted Effect-site Concentration of Propofol (Ceprop) at Certain Time Points
Description: Recording the effect-site concentration of propofol (Ceprop) which showed on target-controlled infusion (TCI) system at loss of consciousness and discontinuation of anesthetics
Time Frame: From anesthesia induction to the patient loss of consciousness, an average of 5 minutes.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Combined Epidural With General Anesthesia | General Anesthesia
Number analyzed (Participants) | 30 | 30
ug/ml | 2.63 (0.38) | 1.97 (0.56)

3. Secondary Outcome: Anesthetics Consumption
Description: Recording the total propofol and reminfentanil consumption during surgery
Time Frame: From anesthesia induction to the end of surgery, an average of 2.5 hours.
Measure: Mean (Standard Deviation); unit: Propofol (mg/Kg.min)
Arm/Group | Combined Epidural With General Anesthesia | General Anesthesia
Number analyzed (Participants) | 30 | 30
Propofol (mg/Kg.min) | 0.11 (0.02) | 0.13 (0.02)

4. Secondary Outcome: Postoperative Exhaust Time
Description: Recording the first postoperative exhaust time by daily follow up
Time Frame: 0-14 days postoperatively
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Combined Epidural With General Anesthesia | General Anesthesia
Number analyzed (Participants) | 30 | 30
hours | 78.0 [58.5 to 110.0] | 85.0 [76.5 to 104.3]

ADVERSE EVENTS:
Time Frame: From anesthesia induction to 6 month after surgery
Arm/Group | Combined Epidural With General Anesthesia | General Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT05124704/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT05124704/SAP_001.pdf